CLINICAL TRIAL: NCT05426395
Title: Single-blinded, Stratified, Multiple Ascending Dose Trial to Assess Pharmacokinetics and Identify Optimal Dose of Vitamin B12 in Pregnancy in Tanzania
Brief Title: Vitamin B12 Dose Escalation Trial in Pregnancy
Acronym: MM4MN-B12
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Principal Investigator, Emily Smith, PI, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MM4MN-B12 2022
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Vitamin B12; Pregnancy
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose 1 (2.6 µg) (Active Comparator): Adding Vitamin B12 at a dose of 2.6 µg
  Interventions: Drug: Vitamin B12 2.6 µg
- Dose 2 (10 µg) (Active Comparator): Adding Vitamin B12 at a dose of 10 µg
  Interventions: Drug: Vitamin B12 10 µg
- Dose 3 (50 µg) (Active Comparator): Adding Vitamin B12 at a dose of 50 µg
  Interventions: Drug: Vitamin B12 50 µg

INTERVENTIONS:
Drug: Vitamin B12 2.6 µg — There are four groups of women (n = 20 total) who will receive B12 dosing once daily, including group 1a (sufficient baseline B12, pregnant), group 1b (sufficient baseline B12, non-pregnant), group 1c (insufficient baseline B12, pregnant), and group 1d (insufficient baseline B12, non-pregnant).
  Arms: Dose 1 (2.6 µg)
Drug: Vitamin B12 10 µg — There are two groups of women (n = 10 total) who will receive B12 dosing once daily, including group 2a (sufficient baseline B12, pregnant) and group 2b (insufficient baseline B12, pregnant).
  Arms: Dose 2 (10 µg)
Drug: Vitamin B12 50 µg — The participants (n = 20 total) will be randomly assigned to receive either a once per day B12 dose or a twice per day B12 dose. The four groups at this dose level include: group 3a (sufficient baseline B12, pregnant, Q12), group 3b (sufficient baseline B12, Q24), group 3c (insufficient baseline B12, pregnant, Q12), group 3d (insufficient baseline B12, Q24).
  Arms: Dose 3 (50 µg)

SUMMARY:
Vitamin B12 is a cofactor for 2 enzymes that have essential functions in pregnancy, both for maternal health and for fetal development. However, there is currently limited data regarding the metabolic fate and optimal dose of supplemental vitamin B12 and its relationship to vitamin B12 status in pregnancy.

This is a single-blinded, stratified, dose-ranging trial of maternal vitamin B12 supplementation during pregnancy that will be conducted at the Ifakara Health Institute Bagamoyo Clinical Trial Unit in Tanzania. The investigators will enroll 40 pregnant women (gestational age 25-28 weeks) and 10 non-pregnant women (comparison group). Participants will be blinded to dosing (2.6, 10, and 50 µg) and supplementation will be given for four weeks.

With this trial, the investigators aim to enhance our understanding of vitamin B12 bioavailability during pregnancy in people with sufficient and insufficient baseline B12 status, identify priority dose regimens of vitamin B12 in pregnancy for investigation in later phase clinical trials to be conducted in populations where vitamin B12 insufficiency or deficiency is common, and identify biomarkers of vitamin B12 intake appropriate for pregnancy.

ELIGIBILITY:
The inclusion criteria for pregnant women are as follows:

* Pregnant female
* Has an estimated gestational age of 25 to 28 weeks at study initiation
* Is between the ages of 18 and 45 years of age
* Lives in the study area and does not plan to travel outside of the study area for the duration of the trial
* Consents to participate in the trial

The exclusion criteria for pregnant women are as follows:

* Known multiple pregnancy (e.g. twins, triplets)
* Has severe anemia (hemoglobin <7 g/dL)
* Has pre-pregnancy or early pregnancy Body Mass Index ≥ 35 kg/m2
* Has a self-reported pre-pregnancy history of type II diabetes mellitus, hypertension, or hypercholesterolemia.
* Has currently diagnosed preeclampsia or eclampsia.
* Has currently diagnosed gestational diabetes.
* Has currently diagnosed renal, liver, autoimmune, or bleeding disorders. The investigators will also assess all women for clinical signs of liver disease including: jaundice or yellowing of skin/sclera/mucosa, right upper quadrant tenderness or pain. All women will be given a liver function test, regardless of clinical signs of liver disease. The tests include: serum Alanine aminotransferase (ALT) and serum Aspartate aminotransferase (AST). Abnormal liver function is defined as the following in this study for women who the investigators screened during the 2nd trimester (25-26 weeks), ALT below 2 or above 33 U/L, or AST below 3 or above 33 U/L; for women screened during the 3rd trimester (27-28 weeks), ALT below 2 or above 25 U/L, or AST below 4 or above 32 U/L (25). Those with liver disease or abnormal liver function will be excluded from the study and referred for treatment.
* Has currently diagnosed congestive heart failure. The investigators will first look for clinical signs of heart failure, and the investigators will focus on the following: i) Fatigue with limitation in performance of normal activities; ii) Coughing, wheezing and breathing difficulty because of lung congestion; iii) Swelling of ankles, feet and legs; and iv) Shortness of breath especially when lying flat. The investigators will only perform lab testing for those who have clinical manifestation, and refer them to appropriate and timely care.
* Has a history of significant gastrointestinal surgeries, such as bariatric surgery, cholecystectomy, or other surgical procedures affecting the stomach, liver, bile ducts and/or small intestine that may disrupt enterohepatic recycling of vitamin B12.
* Has a condition requiring the use of the following medications: H2 blockers, proton pump inhibitors, or prokinetic agents.
* Reports regular use of an over-the-counter, high dose vitamin B12 supplementation. (This criteria does not refer to normal prenatal vitamin supplements which typically include approximately 1 RDA of vitamin B12 or 2.6 ug of vitamin B12. Women using multiple micronutrient supplements, or MMS, are eligible for the study).
* Reports cigarette smoking or tobacco chewing
* Reports heavy alcohol use (>3 drinks per day, or >7 drinks per week)
* Current malaria infection (per rapid diagnostic)
* HIV/AIDS infection (due to potential interaction between first-line antiretroviral dolutegravir and multivitamins that has been shown to decrease dolutegravir exposure by about 33%).
* Has a known allergy to corn or hydroxyethyl starch (HES).

The inclusion criteria for non-pregnant women are as follows:

* Is between the ages of 18 and 45 years of age.
* Lives in the study area and does not plan to travel outside of the study area for the duration of the trial
* Consents to participate in the trial

The exclusion criteria for non-pregnant women are as follows:

* Has severe anemia (hemoglobin <8 g/dL)
* Has Body Mass Index ≥ 35 kg/m2
* Has a self-reported diagnosis of type II diabetes mellitus, hypertension, or hypercholesterolemia.
* Has currently diagnosed renal, liver, autoimmune, or bleeding disorders. The investigators will also assess all women for clinical signs of liver disease including: jaundice or yellowing of skin/sclera/mucosa, right upper quadrant tenderness or pain. Any woman with clinical signs of liver disease will be given a liver function test including: ALT, AST (26,27). Those with liver disease will be excluded from the study and referred for treatment.
* Has currently diagnosed congestive heart failure.
* Has a history of significant gastrointestinal surgeries, such as bariatric surgery, cholecystectomy, or other surgical procedures affecting the stomach, liver, bile ducts and/or small intestine that may disrupt enterohepatic recycling of vitamin B12.
* Has a condition requiring the use of the following medications: H2 blockers, proton pump inhibitors, or prokinetic agents.
* Reports regular use of an over-the-counter, high dose vitamin B12 supplementation.
* Reports cigarette smoking or tobacco chewing
* Reports heavy alcohol use (>3 drinks per day, or >7 drinks per week)
* Current malaria infection (per rapid diagnostic)
* HIV/AIDS infection (due to potential interaction between first-line antiretroviral dolutegravir and multivitamins that has been shown to decrease dolutegravir exposure by about 33%).
* Has a known allergy to corn or hydroxyethyl starch (HES).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessing the steady state pharmacokinetics of B12 upon oral administration in pregnant women. | Over 4 weeks
  The sparse serum vitamin B12 levels measured over 4 weeks at multiple occasions will be used to evaluate the accumulation ratio (steady state B12 level/baseline B12 level) and relative bioavailability between the three doses of B12. The steady state B12 levels will be evaluated descriptively between the three different doses (2.6ug, 10ug and 50ug), different baseline B12 status (sufficient and insufficient), pregnancy status (pregnant and non-pregnant) and other subject specific prognostic factors.
Assessing the steady state pharmacokinetics of B12 upon oral administration in pregnant women. | Over 4 weeks
  The sampling of holotranscobalamin II measured over 4 weeks at multiple occasions will be used to evaluate the absorption and disposition of B12. The mean change from baseline steady state B12 levels in pregnant women will be calculated for the three dose cohorts and the magnitude of difference (fold-change) in mean change from baseline steady state B12 levels between doses will be descriptively compared. Additionally, proportion of subjects who achieved or maintained sufficient B12 status will be assessed for each of the three dose cohorts. A dose with a higher fold difference (from 2.6ug) and higher proportion of women on sufficient status will be identified as a priority B12 dose regimen. The investigators will use metabolomics, proteomics, and genomics to identify novel biomarkers that can more robustly and sensitively reflect vitamin B12 status than conventional markers.
Assessing the steady state pharmacokinetics of B12 upon oral administration in pregnant women. | Over 4 weeks
  The sampling of the ratio of serum B12 to holotranscobalamin measured over 4 weeks at multiple occasions will be used to evaluate the absorption and disposition of B12. The mean change from baseline steady state B12 levels in pregnant women will be calculated for the three dose cohorts and the magnitude of difference (fold-change) in mean change from baseline steady state B12 levels between doses will be descriptively compared. Additionally, proportion of subjects who achieved or maintained sufficient B12 status will be assessed for each of the three dose cohorts. A dose with a higher fold difference (from 2.6ug) and higher proportion of women on sufficient status will be identified as a priority B12 dose regimen. The investigators will use metabolomics, proteomics, and genomics to identify novel biomarkers that can more robustly and sensitively reflect vitamin B12 status than conventional markers.

SECONDARY OUTCOMES:
Assessing serum methylmalonic acid (MMA) | On Day 29
Assessing serum and urinary homocysteine | On Day 29
Assessing hematological response: hemoglobin | On Day 29
Assessing hematological response: hematocrit | On Day 29
Assessing hematological response: erythrocyte count | On Day 29
Assessing hematological response: mean cell volume | On Day 29
Assessing hematological response: reticulocyte number | On Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Ifakara Health Institute Bagamoyo Clinical Trial Unit (BCTU), Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lweno O, Reynolds VS, Barberio MD, Klatt KC, Mugusi S, Gopalakrishnan M, Lukmanji Z, Al-Beity FMA, Ahmadzia HK, Arcot A, Gallagher K, Martin LA, Rahnavard A, Gernand AD, Langevin B, Masanja H, Smith ER. Single-blinded, stratified, dose ranging trial to assess pharmacokinetics and identify optimal dose of vitamin B12 in pregnancy in Tanzania. Gates Open Res. 2025 Sep 17;8:95. doi: 10.12688/gatesopenres.15991.2. eCollection 2024. PMID 41488590